CLINICAL TRIAL: NCT03460249
Title: Office Blood Pressure Measurement With an Automated Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Health Ohio (Other)
Responsible Party: Principal Investigator, Roy Morcos, M.D., Associate Professor of Family and Community Medicine, Mercy Health Ohio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17-015
Record Dates: First submitted 2017-10-18; First posted 2018-03-09 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Blood Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BP table or chair, systolic or diastolic (Active Comparator): record the BP obtained in each patient position
  Interventions: Other: BP measurement
- as above (Active Comparator): as above
  Interventions: Other: BP measurement

INTERVENTIONS:
Other: BP measurement — the BP will be measured in the chair position followed by the table position and also in the reverse sequence

SUMMARY:
The investigators plan to determine if the sequence of blood pressure measurements from the sitting position to the table and vice versa has an impact on the measurements.

DETAILED DESCRIPTION:
The investigators plan to measure blood pressure (BP) in 30 consecutive individuals presenting to the St. Elizabeth Boardman Family Health Center. The sample will include patients presenting for their scheduled appointment. Following informed consent (see attached informed consent form), the participants will be randomly assigned to one of two groups. In group A, the sequence of BP measurements will be table position (TP) followed by recommended chair position (RCP) and then, after a 30-minutes rest, the BP will be measured again in the reverse sequence, RCP then TP. In group B, the sequence will begin with BP measurements in the RCP then TP, followed by 30-minutes rest and then measurements will be repeated in the reverse order. The assignment of participants to groups A and B will be random. The BP will be measured twice in each of the positions described above, according the the accepted standard technique, using a digital blood pressure monitor, the OMRON HEM-907 XL.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the Family Medicine Center age between 18 and 80

Exclusion Criteria:

* Decline to participate for any reason
* Experiencing acute pain or febrile illness
* Pregnant
* Inability to get on the examination table
* Atrial fibrillation, arrhythmia or tachycardia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants whose blood pressures differ with chair to table versus table to chair positioning | 4 months
  Chair to table versus table to chair positional differences in mean systolic and diastolic blood pressures in mm Hg are determined for each participant using an oscillometric device. The percentage of individuals with significant differences in positional blood pressure readings leading to inconsistent blood pressure health status classification will be calculated and reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy Health Youngstown, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No